CLINICAL TRIAL: NCT00146523
Title: An International, Double-Blind, Placebo-Controlled, Study of the Efficacy and Safety of CORLUX™ (Mifepristone) vs. Placebo in the Treatment of Psychotic Symptoms in Patients With Psychotic Major Depression (PMD)
Brief Title: An International Study of the Safety and Tolerability of Corlux for Psychotic Symptoms in Psychotic Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-1073-09
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Major Depressive Disorder
Keywords: Psychotic Major Depression; PMD; Depression; Major Depression; Psychosis
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Psychotic Disorders | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- mifepristone 600 mg (Experimental)
  Interventions: Drug: Mifepristone
- matching placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mifepristone
  Arms: mifepristone 600 mg
Drug: placebo
  Arms: matching placebo

SUMMARY:
Corlux (mifepristone) is a new medication that modulates the body's use of a hormone called cortisol. Under normal conditions, cortisol and other hormones are created by the body in response to physical and emotional stress, triggering a healthy stress response. People who suffer from psychotic major depression may have unusually high levels of cortisol circulating within them or abnormal patterns of cortisol levels, overloading the stress response mechanism and causing symptoms of psychosis such as delusional thoughts or hallucinations. If Corlux can keep the body's cortisol receptors from being overloaded, the stress response system may return to normal function, which may result in improvement of symptoms. The purpose of this 56 day study is to learn the safety and effectiveness of Corlux in patients who have been diagnosed with psychotic major depression (PMD).

ELIGIBILITY:
Inclusion Criteria:

* Are 18 to 75 years of age
* Have a diagnosis of major depressive disorder with psychotic features (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition [DSM IV] 296.24 or 296.34)
* Are able to provide written informed consent.

Exclusion Criteria:

* Have a major medical problem
* Have previously participated in a Corlux (C-1073, mifepristone) clinical trial
* Have a history of an allergic reaction to Corlux (C-1073, mifepristone).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2005-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The change in a measure of psychosis | screening and on Days 0, 7, 14, 28, 42, and 56

SECONDARY OUTCOMES:
The change in a measure of depression | screening and on Days 0, 7, 14, 28, 42, and 56

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Beebe, PhD, Study Director — Corcept Therapeutics
Locations (19):
- Bulgaria (5):
  - Georgy Koychev M.D., Sofia
  - Luchezar G Hranov M.D., Sofia
  - Svetlozar H Haralanov Ph.D., Sofia
  - Vihra Milanova M.D., Sofia
  - Georgi Popov M.D., Varna
- Croatia (6):
  - Pavo Filakovic M.D./Ph.D., Osijek
  - Ljiljana Moro M.D./Ph.D., Rijeka
  - Goran Dodig M.D./Ph.D., Split
  - Dubravka Kocijan-Hercigonja M.D., Zagreb
  - Miro Jakovljevic M.D., Zagreb
  - Vera Folnegovic-Smalc M.D./Ph.D., Zagreb
- Romania (2):
  - Mihai Dumitru Gheorge, Bucharest
  - Aurel Nirestean M.D./Ph.D., Târgu Mureş
- Serbia and Montenegro (6):
  - Ivana Timotijevic M.D., Belgrade
  - Jelena Martinovic M.D., Belgrade
  - Vladimir Diligenski M.D., Belgrade
  - Vladimir Paunovic M.D., Belgrade
  - Dragana Ignjatovic-Ristic M.D., Kragujevac
  - Ratomir Lisulov M.D., Novi Sad

REFERENCES:
- [Background] Belanoff JK, Rothschild AJ, Cassidy F, DeBattista C, Baulieu EE, Schold C, Schatzberg AF. An open label trial of C-1073 (mifepristone) for psychotic major depression. Biol Psychiatry. 2002 Sep 1;52(5):386-92. doi: 10.1016/s0006-3223(02)01432-4. PMID 12242054
- [Background] Brogden RN, Goa KL, Faulds D. Mifepristone. A review of its pharmacodynamic and pharmacokinetic properties, and therapeutic potential. Drugs. 1993 Mar;45(3):384-409. doi: 10.2165/00003495-199345030-00007. PMID 7682909
- [Background] Belanoff JK, Flores BH, Kalezhan M, Sund B, Schatzberg AF. Rapid reversal of psychotic depression using mifepristone. J Clin Psychopharmacol. 2001 Oct;21(5):516-21. doi: 10.1097/00004714-200110000-00009. PMID 11593077
- [Derived] Block TS, Kushner H, Kalin N, Nelson C, Belanoff J, Schatzberg A. Combined Analysis of Mifepristone for Psychotic Depression: Plasma Levels Associated With Clinical Response. Biol Psychiatry. 2018 Jul 1;84(1):46-54. doi: 10.1016/j.biopsych.2018.01.008. Epub 2018 Jan 31. PMID 29523415
- See also: Corcept Therapeutics — http://www.corcept.com